CLINICAL TRIAL: NCT00726401
Title: A Randomized, Double-blind, Placebo-controlled Study on the Effect of CVT-E002 in Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afexa Life Sciences Inc (Industry)
Responsible Party: Dr. Jacqueline Shan, Afexa Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT-E002-2007-2
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Allergies; Nasal; Congestion; Sneezing; Pruritus; Teary; Eyes
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity; Sneezing; Pruritus | interventions — COLD-fX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: COLD-fX
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COLD-fX — 200mg BID for 4 weeks
  Other Names: CVT-E002
  Arms: 1
Drug: Placebo — 200mg BID for 4 weeks
  Arms: 2

SUMMARY:
You are being asked to take part in a research study of COLD-fX, a product designed to boost the immune system. COLD-fX is an extract from the roots of North American ginseng and it may offer some benefit to people with seasonal allergies.

The purpose of the present study is to find out how effective and safe COLD-fX is in improving quality of life and reducing symptoms of seasonal allergies such as hay fever. COLD-fX is not yet approved for treatment of seasonal allergies. We are seeking to enroll 200 participants in the Capital Health region.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study will be carried out to establish the effects of CVT-E002 200 mg twice daily for 4 weeks in patients with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals of both genders aged 12 - 75 years
2. Documented clinical history of seasonal allergic rhinitis for at least 2 years with exacerbations during the study season; and exhibit a positive skin-prick test (wheal diameter at least 3 mm greater than saline control) to one of the regional allergens active during the study season
3. Determined by the investigators that well-controlled mild to moderate asthmatics will not be excluded
4. Daytime nasal symptoms of at least mild-to-moderate severity (cumulative score of at least 42 over a 7-day run-in period)
5. Women of child bearing capacity who agree to use an acceptable form of birth control during the trial (i.e., oral contraception, reliable use of a double-barrier method (e.g., condom and diaphragm, condom and foam, condom and sponge), IUD, or tubal ligation)
6. Willing to adhere to the requirements of the protocol, including availability for follow-up visits
7. Willing and able to sign written informed consent

Exclusion Criteria:

1. Medical conditions:

   * Perennial rhinitis with little or no seasonal flare-ups
   * Rhinitis medicamentosa
   * Non-allergic rhinitis
   * Nasal polyps
   * Severe asthma that is poorly controlled
   * Active tuberculosis
   * Cystic fibrosis
   * Upper respiratory tract infection within the preceding 4 weeks
   * Significant other pulmonary disorders
   * Any ongoing allergen immunotherapy during study or for 6 months prior
   * HIV/AIDS
   * Malignancy (under active observation or treatment)
   * Unstable cardiovascular disease (physician visit or hospitalization for unstable cardiovascular disease in the last 6 months)
   * Renal abnormalities (serum creatinine known to be > 200 mmol/l)
   * Acute or active chronic liver disease
   * Diabetes
   * Neurological or psychiatric disease (progressive or currently under treatment)
   * Bleeding disorders
   * Major surgery in the last 6 months or planned surgery over the course of the study
   * Other serious medical conditions
2. Medications:

   * Medications for allergic rhinitis/conjunctivitis, including: antihistamines; oral, parenteral, nasal, and ophthalmic corticosteroids; cromolyn sodium; nedocromil; and intranasal anticholinergics (If the participants agree to stop taking these products prior to study entry and for the duration of the study, they can participate in the study.)
   * Oral or long-acting b-agonists, theophylline, and leukotriene modifiers
   * Medications that can affect nasal or ocular symptoms, including decongestants and anti-inflammatory drugs
   * Allergic rhinitis rescue medications
   * Use of immunosuppressants
   * Hormone replacement therapy
   * Phenelzine
   * Pentobarbital
   * Haloperidol
   * Warfarin
   * Heparin
   * Any other natural health products or dietary supplements, with the exception of vitamins and minerals with dose of > 600 mg/day of vitamin E and containing no vitamin K. Natural health products or dietary supplements include products such as, but not limited to, Echinacea, Ginseng (beverages, foods, extracts, capsules, or tablets), St. John's Wort, Gingko, Glucosamine, Fish Oil supplements, Evening Primrose Oil, Green Tea or other herbal products consumed in the form of a pill or capsule. (If the participants agree to stop taking these products prior to study entry and for the duration of the study, they can participate in the study.)
3. Daily smokers (> 25 cigarettes per day)
4. History of alcohol/drug abuse
5. Suspected substance abuse or dependence active within the preceding 4 weeks
6. Pregnant or breast-feeding women
7. Allergy to ginseng, microcrystalline cellulose, or gelatin

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Preliminary estimates of treatment effect of CVT-E002 in improving quality of life and reducing symptoms | 4 weeks

SECONDARY OUTCOMES:
Safety and tolerability of CVT-E002 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Predy, FFCPC, Principal Investigator — Capital Health, Canada
Locations (4):
- Canada (4):
  - Capital Health, Edmonton, Alberta
  - McMaster University Medical Centre, Hamilton, Ontario
  - Melimar Allergy Laboratory, Toronto, Ontario
  - JDM Research, Toronto, Ontario